CLINICAL TRIAL: NCT02039557
Title: Long Term Follow Up for Patients Who Have Received Allogeneic Stem Cell Transplantation of NiCord®/CordIn™, Umbilical Cord Blood-derived Ex Vivo Expanded Stem and Progenitor Cells
Brief Title: Long Term Follow Up Protocol for NiCord®/CordIn™ (Omidubicel) Patients
Status: Completed | Type: Observational
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: GC P# 04.01.020/030
Record Dates: First submitted 2014-01-13; First posted 2014-01-17 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Patients Transplanted With NiCord/CordIn (Omidubicel)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NiCord®/CordIn™ (omidubicel) transplanted: Anyone who signed the consent for this study received a NiCord®/CordIn™ (omidubicel) infusion as part of a GC clinical interventional study, and completed the interventional study Day 365 status assessment.
  Interventions: Genetic: NiCord®/CordIn™ (omidubicel)

INTERVENTIONS:
Genetic: NiCord®/CordIn™ (omidubicel)

SUMMARY:
This is an observational study that will monitor clinical outcomes of patients who have received a NiCord®/CordIn™ (omidubicel) transplant as part of a GC clinical interventional study and meet the eligibility criteria for this Long Term Follow Up study.

ELIGIBILITY:
Inclusion Criteria

* Anyone who has received a NiCord®/CordIn™ (omidubicel) transplant, completed study specific follow up, and has signed the consent for this study.

Exclusion Criteria

* None

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NiCord® (ages 12-65)/CordIn™ (ages 2-25) (omidubicel) transplanted patients
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
long term sustained chimerism of NiCord®/CordIn™ (omidubicel) transplantation | 5 years

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt, Nashville, Tennessee
- University Medical Center Utrecht, Utrecht, Netherlands
- Singapore (2):
  - National University Cancer Institute, Singapore
  - Singapore General Hospital, Singapore
- Spain (2):
  - University Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario La Fe, Valencia